CLINICAL TRIAL: NCT06078969
Title: The Efficacy of Oral Prednisone in Treating Langerhans Cell Histiocytosis of Bone in Childhood and Adolescence: A Multi-center, Open-label, Randomized-controlled, Phase II Study
Brief Title: Oral Prednisone in Treating LCH of Bone in Childhood and Adolescence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Peking University Third Hospital (Other); National Sun Yat-sen University (Other); Beijing Children's Hospital (Other); Henan Cancer Hospital (Other Government); Tianjin Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Second Hospital of Jilin University (Other); Peking University People's Hospital (Other); Jinling Hospital, China (Other); The First Affiliated Hospital of Nanchang University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Jianru Xiao, Professor, Chief Surgeon, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023SL049
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Langerhans Cell Histiocytosis of Bone
Keywords: Langerhans cell histiocytosis; Bone; Single-system; Children; Adolescents
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: If the diseae progression in the control group is confirmed, the patient is allowed to transferred to the test group (Oral prednisone).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral prednisone (Experimental): Oral prednisone, 0.5mg/kg/day, first 5 days/month, 6months
  Interventions: Drug: Prednisone
- Regular observation (No Intervention): Regular observation and follow up without medication

INTERVENTIONS:
Drug: Prednisone — For the experimental group, the patient will be administrated oral prednisone (0.5mg/kg/day, first 5 days per month, 6 months)
  Arms: Oral prednisone

SUMMARY:
Langerhans cell histiocytosis (LCH) of bone is a benign-tumor-like osteolytic lesion in childhood and adolescence, which is characterized by the aberrant activation of antigen presenting cells. Rather than the multi-system involvements of LCH, no standard or widely-accepted therapeutic regimens were established for LCH of bone. In the previous clinical practice, several LCH patients obtained remarkable pain relief after taking prednisone. Therefore, the investigators aim to conducting a multi-center, open-labelled, randomized-controlled, Phase II study to investigate the efficacy and safety of oral prednisone in treating LCH of bone in children and adolescents. The enrolled patients will be randomly recruited to the following groups: (1) Oral prednisone [Test group); (2) Regular observation [Control group].

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of Langerhans cell histiocytosis (LCH) of bone;
* Single-system involvement (skeletal system);
* No need of surgical intervention;
* Must be able to swallow tablets;
* Signing informed consent form.

Exclusion Criteria:

* Multi-system involvements (≥2 systems, including bone, liver, spleen, hematologic system, central nerve system);
* Need of surgical intervention (e.g. pathological fracture and/or spinal cord compression)
* Glucocorticoid allergy;
* Immunodeficiency;
* Severe infection;
* Insulin dependent/independent Diabetes;
* Having taken glucocorticoid in the past two weeks;
* Not capable of swallowing tablets;
* Without signed informed consent inform.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Any evidence proving the disease progression

SECONDARY OUTCOMES:
Local control rate | 2 years
  radiological examinations of local lesion status
Pain relief | 2 years
  The Visual Analogue Scale (Minimum: 0; Maximum: 10 scores), is used to evaluate the degree of pain relief. The higher scores mean a worse outcome.
Adverse effect rate | 2 years
  side effects related to the prednisone

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 1 year

REFERENCES:
- [Background] Stull MA, Kransdorf MJ, Devaney KO. Langerhans cell histiocytosis of bone. Radiographics. 1992 Jul;12(4):801-23. doi: 10.1148/radiographics.12.4.1636041.
- [Background] Gadner H, Minkov M, Grois N, Potschger U, Thiem E, Arico M, Astigarraga I, Braier J, Donadieu J, Henter JI, Janka-Schaub G, McClain KL, Weitzman S, Windebank K, Ladisch S; Histiocyte Society. Therapy prolongation improves outcome in multisystem Langerhans cell histiocytosis. Blood. 2013 Jun 20;121(25):5006-14. doi: 10.1182/blood-2012-09-455774. Epub 2013 Apr 15. PMID 23589673
- [Background] Mitchell P, Ezeokoli EU, Borici N, Schleh E, Montgomery N. Treatment and Outcomes of Unifocal and Multifocal Osseous Pelvic Langerhans Cell Histiocytosis Lesions in a Pediatric Population. Cureus. 2022 Aug 27;14(8):e28470. doi: 10.7759/cureus.28470. eCollection 2022 Aug. PMID 36176854
- [Background] Baptista AM, Camargo AF, de Camargo OP, Odone Filho V, Cassone AE. Does adjunctive chemotherapy reduce remission rates compared to cortisone alone in unifocal or multifocal histiocytosis of bone? Clin Orthop Relat Res. 2012 Mar;470(3):663-9. doi: 10.1007/s11999-011-2162-x. PMID 22052526
- [Background] Zhong N, Xu W, Meng T, Yang X, Yan W, Xiao J. The surgical strategy for eosinophilic granuloma of the pediatric cervical spine complicated with neurologic deficit and/or spinal instability. World J Surg Oncol. 2016 Dec 7;14(1):301. doi: 10.1186/s12957-016-1063-6. PMID 27923375
- [Background] Tang X, Gao J, Ma ZG, Guo X, Li Q, Wan Z, Sun JJ. Clinical and prognostic characteristics of 95 cases of Langerhans cell histiocytosis in children: a single-institute experience from 2013 to 2020. Ann Med. 2021 Dec;53(1):1537-1546. doi: 10.1080/07853890.2021.1966085. PMID 34459688